CLINICAL TRIAL: NCT02045277
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Vehicle Controlled Clinical Study to Assess the Safety and Efficacy of IDP 118 in the Treatment of Plaque Psoriasis
Brief Title: Safety and Efficacy of IDP 118 in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-118A-201
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Transcriptional Coactivator with PDZ-Binding Motif Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDP-118 Lotion (Experimental): halobetasol propionate [HP], tazarotene [Taz]
  Interventions: Drug: IDP-118 Lotion
- IDP-118 Monad HP Lotion (Active Comparator): HP
  Interventions: Drug: IDP-118 Monad HP Lotion
- IDP-118 Monad Taz Lotion (Active Comparator): Taz
  Interventions: Drug: IDP-118 Monad Taz Lotion
- IDP-118 Vehicle Lotion (Active Comparator): Vehicle
  Interventions: Drug: IDP-118 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-118 Lotion — Lotion
  Other Names: Lotion
  Arms: IDP-118 Lotion
Drug: IDP-118 Monad HP Lotion — Active Comparator
  Other Names: HP
  Arms: IDP-118 Monad HP Lotion
Drug: IDP-118 Monad Taz Lotion — Active Comparator
  Other Names: Taz
  Arms: IDP-118 Monad Taz Lotion
Drug: IDP-118 Vehicle Lotion — Vehicle
  Other Names: Vehicle
  Arms: IDP-118 Vehicle Lotion

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of a topical lotion

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and efficacy of a topical lotion when applied once daily to adult subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, of any race, at least 18 years of age (inclusive).
* Freely provides both verbal and written informed consent.
* Has an area of plaque psoriasis appropriate for topical treatment that covers a BSA of at least 3%, but no more than 12%. The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this calculation.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Has a clinical diagnosis of psoriasis at the Baseline visit with an IGA score of 3 or 4. (The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this assessment, if psoriasis is present).

Key Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or pustular psoriasis, as determined by the investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the investigator.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half lives (whichever is longer) prior to the Baseline visit, or is concurrently participating in another clinical study with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu J Alexander, Study Director — Valeant Pharmaceuticals
Locations (18):
- United States (18):
  - Valeant Site 13, Encino, California
  - Valeant Site 11, San Diego, California
  - Valeant Site 15, Santa Rosa, California
  - Valeant Site 10, Augusta, Georgia
  - Valeant Site 09, Newnan, Georgia
  - Valeant Site 08, Louisville, Kentucky
  - Valeant Site 04, Rockville, Maryland
  - Valeant Site 14, Clinton Township, Michigan
  - Valeant Site 07, Fridley, Minnesota
  - Valeant Site 01, East Windsor, New Jersey
  - Valeant Site 03, New York, New York
  - Valeant Site 17, Rochester, New York
  - Valeant Site 02, High Point, North Carolina
  - Valeant Site 05, Austin, Texas
  - Valeant Site 06, College Station, Texas
  - Valeant Site 16, Salt Lake City, Utah
  - Valeant Site 18, Lynchburg, Virginia
  - Valeant Site 12, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-118 Lotion | IDP-118 Monad HP Lotion | IDP-118 Monad Taz Lotion | IDP-118 Vehicle Lotion
Started | 59 | 63 | 59 | 31
Completed | 55 | 62 | 47 | 29
Not Completed | 4 | 1 | 12 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-118 Lotion | IDP-118 Monad HP Lotion | IDP-118 Monad Taz Lotion | IDP-118 Vehicle Lotion | Total
Number analyzed (Participants) | 59 | 63 | 59 | 31 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (13.70) | 54.2 (11.52) | 55.7 (13.10) | 52.4 (16.11) | 52.66 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 19 | 12 | 79
  Male | 35 | 39 | 40 | 19 | 133

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success of a 2-Grade IGA Score Improvement From Baseline and an IGA Score of Clear or Almost Clear at Week 8
Description: Treatment success defined as at least a 2-grade improvement from Baseline in the IGA score and an IGA score equating to "clear" or "almost clear" at Week 8. The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe).
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | IDP-118 Lotion | IDP-118 Monad HP Lotion | IDP-118 Monad Taz Lotion | IDP-118 Vehicle Lotion
Number analyzed (Participants) | 59 | 63 | 59 | 31
percentage of participants | 52.5 | 33.3 | 18.6 | 9.7

2. Primary Outcome: Percentage of Participants With Treatment Success of a 2-Grade IGA Score Improvement From Baseline and an IGA Score of Clear or Almost Clear at Weeks 2, 4, 6, and 12
Description: Treatment success defined as at least a 2-grade improvement from Baseline in the Investigator's Global Assessment (IGA) score and an IGA score equating to "clear" or "almost clear" at Weeks 2, 4, 6, and 12. The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe).
Time Frame: Weeks 2, 4, 6, and 12 (4-week follow-up)
Population: The number of participants with IGA results at each visit were utilized in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | IDP-118 Lotion | IDP-118 Monad HP Lotion | IDP-118 Monad Taz Lotion | IDP-118 Vehicle Lotion
Number analyzed (Participants) | 59 | 63 | 59 | 31
percentage of participants
  Week 2 | 11.9 | 4.8 | 1.7 | 0
  Week 4 | 25.4 | 17.5 | 1.7 | 6.5
  Week 6 | 32.2 | 25.4 | 15.3 | 3.2
  Week 12: number analyzed (Participants) | 55 | 62 | 47 | 29
  Week 12 | 38.2 | 21.0 | 12.8 | 6.9

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were collected from participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-Baseline safety assessment (Safety Population).
Arm/Group | IDP-118 Lotion | IDP-118 Monad HP Lotion | IDP-118 Monad Taz Lotion | IDP-118 Vehicle Lotion
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/62 | 1/58 | 2/31
Other Adverse Events (participants affected / at risk) | 7/59 | 0/62 | 9/58 | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=59) | IDP-118 Monad HP Lotion (N=62) | IDP-118 Monad Taz Lotion (N=58) | IDP-118 Vehicle Lotion (N=31)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Hernia obstructive (General disorders) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=59) | IDP-118 Monad HP Lotion (N=62) | IDP-118 Monad Taz Lotion (N=58) | IDP-118 Vehicle Lotion (N=31)
Application site erythema (General disorders) | 1 | 0 | 3 | 0
Application site pain (General disorders) | 2 | 0 | 5 | 1
Application site pruritus (General disorders) | 2 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 3 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.